CLINICAL TRIAL: NCT02783534
Title: Manual Acupuncture vs Sham Acupuncture and Usual Care for the Prevention of Primary Dysmenorrhea: A Multicenter, Randomized, Controlled, Clinical Trial
Brief Title: Manual Acupuncture for Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Hubei College of Traditional Chinese Medicine (Other); Hubei Hospital of Traditional Chinese Medicine (Other); Wuhan Integrated Traditional Chinese and Western Medicine Hospital (Other); University Hospital of Huang Jia Lake Campus, Hubei University of Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Wei Wang, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201403RCTPD
Record Dates: First submitted 2016-05-05; First posted 2016-05-26 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Primary Dysmenorrhea
Keywords: Acupuncture; Primary Dysmenorrhea; Randomized Controlled Trial; Placebo Effect

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Verum acupuncture (Experimental): Participants will receive verum acupuncture plus usual care. Participants will receive acupuncture treatment start from the 5th or 7th day before the estimated first day of menstrual cycle, and for each cycle, participants will receive one session of treatment each day for 5 consecutive days, totally be treated with 15 sessions.Verum needles will be inserted into the skin and manipulated manually until deqi occurs. The needles are retained for 30 min in each session. During the treatment, the acupuncturist inquires the patient about deqi sensations and manipulates the needles to maintain the intensity of deqi. Participants will receive the same usual care as those in the usual care group.
  Interventions: Device: Verum acupuncture; Behavioral: Usual care
- Sham acupuncture (Sham Comparator): Participants will receive sham acupuncture plus usual care. The Streitberger placebo needle will be placed at non-acupuncture points which are distant from the meridian parts and not located on the same neuromuscular segments as the prescribed points used in the VA group, so as to minimize any therapeutic and segmental effects. The same acupuncture schedule as that in the verum acupuncture group will be applied. The needles are retained for 30 min in each session. During the treatment, the acupuncturist inquires the patient about deqi sensations and pretends to manipulate the needles but deqi is not sought.Participants will receive the same usual care as those in the usual care group.
  Interventions: Device: Sham acupuncture; Behavioral: Usual care
- Usual care (Placebo Comparator): Participants will not receive acupuncture treatment besides health education as a control group.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Device: Verum acupuncture — Participants allocated to VA group will receive traditional acupuncture treatment on the "Guanyuan"(RN 4), bilateral "Sanyinjiao"(SP 6), bilateral "Zigong"(EX-CA1), bilateral "Xuehai"(SP 10). Additional points will be chosen according to TCM syndrome differentiation constitution of patients. If patients with deficient syndrome, bilateral "Zusanli" (ST 36) will be included. If patients with sufficiency syndrome, bilateral "Diji" (SP 8) will be included. The NO.16 special type of acupuncture needle (0.30 x 30 mm) produced by German asia-med company will be applied.The needles will be inserted into the skin of acupuncture points and manipulated manually by using the techniques such as lifting, thrusting, and twirling, until the internal compound sensation known as deqi.
  Arms: Verum acupuncture
Device: Sham acupuncture — We use a non-insertive sham control produced by Asia-med Company in Germany-the streitberger placebo-needle. Sham points are described as follows: 1) 5 inch lateral to the seventh thoracic spine; 2) 5 inch lateral to the eighth thoracic spine; 3) 5 inch lateral to the ninth thoracic spine; and 4) 5 inch lateral to the tenth thoracic spine.
  Arms: Sham acupuncture
Behavioral: Usual care — Patients in usual care group will not receive acupuncture treatment but enhance usual care by providing them with detailed information via propaganda booklets or the internet in the form of health education.

SUMMARY:
Primary dysmenorrhea (PD) is a common complaint in menstruating women. Although nonsteroidal anti-inflammatory drug is an effective treatment, there are concerns about serious adverse events. Complementary therapies, including acupuncture, are commonly used for PD. Acupuncture has a low risk of adverse effects, while the evidence for the effectiveness of acupuncture in treating PD is inconclusive. Deqi and psychological factors are core concepts in acupuncture theory, but they have been largely neglected in primary dysmenorrhea clinical reports. The objective of this trail is to assess the clinical efficacy of acupuncture in the prevention of PD and investigate what factors will affect the efficacy of acupuncture.The results of this trial will significantly add to the current body of evidence on the role of acupuncture for PD. If found to be effective and safe, acupuncture will be a valuable treatment option in the prevention of PD. In additional, results from this trial will identify what factors will affect the efficacy of acupuncture.

DETAILED DESCRIPTION:
This is a multicenter, single blind, randomized controlled, three-arm, large-scale clinical trial. We will recruit 300 PD women who meet diagnostic criteria for PD established in 2005 from Canada gynaecology and obstetrics association. Exclusion criteria include illiteracy, breast feeding women, pregnancy women, serious systemic disease, mental patient, and acupuncture experience. Eligible women will be randomly assigned to verum acupuncture group, sham acupuncture group and usual care group. Participants in the verum acupuncture group will receive traditional acupuncture treatment and will be treated with ture needles, While Participants in the sham acupuncture group will be treated with sham acupuncture with non-insertive needles at non-acupuncture points. Acupuncture treatment will start from the 5th or 7th day before the estimated first day of menstrual cycle, and for each cycle, participants will receive one session of treatment each day for 5 consecutive days (a treatment course), totally for 15 sessions and 3 treatment courses. Participants in the usual care group will not receive treatment besides health education as a control group. This trail will be composed of a one-menstrual cycle baseline, three-menstrual cycle treatment (cycle 1 to 3), and three-menstrual cycle follow-up period (cycle 4-6). The primary outcome measure is the change of Cox Menstrual Symptom Scale (CMSS) in a menstrual cycle compared to baseline. Secondary outcome measures include Visual Analogue Scale (VAS), McGill pain questionnaire (SF-MPQ), Pittsburgh sleep quality index (PSQI), and intake of acute medication. Psychological outcome measures are Beck Depression Rating Scale (BDI), Beck Anxiety Inventory (BAI), NEO Five-Factor Inventory (NEO-FFI), the Doctor-Patient Relationship Scale (PDRQ), the Difficult Doctor-Patient Relationship Questionnaire (DDPRQ), and Expectations for interventions assessed by acupuncture expectancy scale (AES). Deqi sensation will be measured by MGH Acupuncture Sensation Scale (MASS).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with PD according to the primary dysmenorrhea established by Canadian Institute of Obstetrics and gynecology in 2005;
2. Aged from 15 to 40 years, have not given birth, and have a history of regular menstrual cycles (28 days±7 days);
3. Pain of intensity is moderate varying from 40 to 80 on the visual analogue scale (VAS), and lasting at least 6 months;
4. Able to complete the baseline dysmenorrhea diary;
5. Able to sign an informed consent

Exclusion Criteria:

1. Secondary dysmenorrhea caused by endometriosis, pelvic inflammation, myomas of uterus or other gynecological problems confirmed by type-B ultrasound exam by gynecologists;
2. Have a history of pelvic or abdominal surgery, or applying oral contraceptives or intrauterine devices;
3. Combined with uncontrolled diagnosed psychiatric disorders such as severe anxiety and depression, or severe systemic diseases affecting the implementation of treatment programs;
4. Taking analgesics such as NSAIDs or having received any other treatment for PD three months prior to enrollment;
5. Women in lactation, pregnant women, or those with plans to get pregnant during any period of the trial;
6. Have experience of acupuncture;
7. Illiterate, or patients unable to read and understand scales.

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-08-02 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Change of Cox Menstrual Symptom Scale (CMSS) in a menstrual cycle compared to baseline. | At baseline (one menstrual cycle/one month before randomization), the first，second, third, fourth, fifth, and sixth month after randomization.

SECONDARY OUTCOMES:
Change of Visual Analogue Scale (VAS) in a menstrual cycle compared to baseline. | At baseline (one menstrual cycle/one month before randomization), the first，second, third, fourth, fifth, and sixth month after randomization.
Change of McGill pain questionnaire (SF-MPQ) in a menstrual cycle compared to baseline. | At baseline (one menstrual cycle/one month before randomization), the first，second, third, fourth, fifth, and sixth month after randomization.
Change of Pittsburgh sleep quality index (PSQI) in a menstrual cycle compared to baseline. | At baseline (one menstrual cycle/one month before randomization), the first，second, third, fourth, fifth, and sixth month after randomization.
Change of the dose of intake of acute medication in a menstrual cycle compared to baseline. | At baseline (one menstrual cycle/one month before randomization), the first，second, third, fourth, fifth, and sixth month after randomization.

OTHER OUTCOMES:
Chinese version of Massachusetts General Hospital Acupuncture Sensation Scale | From date of the first session of treatment until date of the fifteenth session of treatment, assessed up to 75 days.
Change in Beck Depression Inventory II (BDI- II) compared to baseline. | At baseline (one menstrual cycle/one month before randomization), at the third month after randomization, and at the sixth month after randomization.
Change in Beck Anxiety Inventory (BAI) compared to baseline. | At baseline (one menstrual cycle/one month before randomization), at the third month after randomization, and at the sixth month after randomization.
60-item NEO Personality Inventory-Short Form (NEO-FFI) | At baseline (one menstrual cycle/one month before randomization) only once.
Patient-Doctor Relationship Questionnaire (PDRQ-9). | At baseline (one menstrual cycle/one month before randomization), at the third month after randomization, and at the sixth month after randomization.
Acupuncture expectancy scale | Before the first session of treatment, at the end of the third session of treatment (on day 3), and at the end of the fifteenth session of treatment (up to 75 days).
Chinese medicine constitution questionnaire | At baseline (one menstrual cycle/one month before randomization), at the third month after randomization, and at the sixth month after randomization.
Difficult Doctor-Patient Relationship Questionnaire (DDPRQ-10). | At baseline (one menstrual cycle/one month before randomization), at the third month after randomization, and at the sixth month after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Department of Neurology of Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu L, Liu S, Zheng C, Liu W, Wang H, Liang F, Lu W, Xu S, Wang W. Manual acupuncture versus sham acupuncture and usual care for the prevention of primary dysmenorrhea (PD): study protocol for a randomized controlled trial. Trials. 2020 Sep 29;21(1):818. doi: 10.1186/s13063-020-04720-5. PMID 32993752